CLINICAL TRIAL: NCT02638519
Title: Hyperpolarized Xenon-129 Functional Magnetic Resonance Imaging of Healthy Volunteers and Participants With Alzheimer's Disease
Brief Title: HP Xenon-129 fMRI of Healthy Volunteers and Participants With Alzheimer's Disease
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Unable to reach the target enrollment of 40 participants with Alzheimer's disease.
Sponsor: Thunder Bay Regional Health Research Institute (Other)
Collaborators: Lakehead University (Other); Thunder Bay Regional Health Sciences Centre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: RP-307-08312015
Record Dates: First submitted 2015-12-03; First posted 2015-12-23 (Estimated); Last update posted 2024-10-15 (Actual); Status verified 2024-08

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Healthy Volunteers (Other): Healthy volunteers will inhale NeuroXene using various breathing methods. The CMRS 1H-129Xe dual-tuned quadrature head coil will be used to acquire MRI images of the human brain after inhalation of NeuroXene. The coil permits the acquisition of both conventional proton and HP xenon gas images. Two types of MRI scans will be performed: Traditional proton fMRI and Hyperpolarized Xenon-129 fMRI. The order of scans will be randomized to account for bias caused by scan order.
  Interventions: Other: Traditional Proton fMRI; Other: Hyperpolarized Xenon-129 fMRI; Drug: Hyperpolarized Xenon-129; Device: 1H-129Xe Dual-Tuned Quadrature Head Coil
- Alzheimer's Disease Participants (Other): Alzheimer's disease participants will inhale NeuroXene using various breathing methods. The CMRS 1H-129Xe dual-tuned quadrature head coil will be used to acquire MRI images of the human brain after inhalation of NeuroXene. The coil permits the acquisition of both conventional proton and HP xenon gas images. Two types of MRI scans will be performed: Traditional proton fMRI and Hyperpolarized Xenon-129 fMRI. The order of scans will be randomized to account for bias caused by scan order.
  Interventions: Other: Traditional Proton fMRI; Other: Hyperpolarized Xenon-129 fMRI; Drug: Hyperpolarized Xenon-129; Device: 1H-129Xe Dual-Tuned Quadrature Head Coil

INTERVENTIONS:
Other: Traditional Proton fMRI — Conventional proton fMRI will be performed. During the functional imaging acquisitions, the participant will be asked by the research team to perform simple tasks. These tasks will be completed while the participant breathes air (normal breathing).
Other: Hyperpolarized Xenon-129 fMRI — HP 129Xe fMRI data will be acquired from all participants. Hyperpolarized xenon (NeuroXene) is expected to produce images that provide more clinically relevant information than traditional proton scans. Simple tasks will be performed by participants while breathing NeuroXene according to several inhalation procedures.
  Other Names: HP 129Xe fMRI
Drug: Hyperpolarized Xenon-129 — Participants will be asked to inhale specified amounts of NeuroXene according to several inhalation procedures. NeuroXene is the trade name for hyperpolarization of xenon-129 balanced with oxygen and nitrogen using a Xemed LLC polarizer. Hyperpolarization does not change the chemical or physical properties of xenon gas.
  Other Names: NeuroXene
Device: 1H-129Xe Dual-Tuned Quadrature Head Coil — A 1H-129Xe dual-tuned quadrature head coil (Clinical MR Solutions, LLC) will be used in this study. The RF coil will be used to acquire MRI images of the human brain after inhalation of hyperpolarized xenon-129 gas, and permits the acquisition of both conventional proton and HP xenon gas images.

SUMMARY:
This study involves imaging participants' brains using MRI. The goal is to develop a high-resolution, high-sensitivity imaging tool, hyperpolarized xenon functional brain magnetic resonance imaging, which can provide more sensitive measurement of brain function, facilitating the development of drugs for more successful treatment of Alzheimer's disease.

DETAILED DESCRIPTION:
The described study is a pilot study in which the investigators aim to develop an enhanced sensitivity tool for assessment of neural function. Participation involves at least two study visits no longer than three hours in length each. During visit 1, informed consent and screening for eligibility will take place. During visit 2, fMRI scanning will take place in which participants will complete simple tasks. Two types of MRI scans will be performed: traditional proton fMRI and hyperpolarized xenon-129 fMRI (HP 129Xe fMRI) scans. The trade name for xenon-129 hyperpolarized with a Xemed LLC polarizer is NeuroXene.

Participants will be placed in the 3T MRI at the Thunder Bay Regional Research Institute with a Clinical MR Solutions (CMRS) Dual Brain Coil that fits over their head like a helmet. Several inhalation procedures will be performed by participants when breathing NeuroXene from a tube in the scanner. Preparation and administration of NeuroXene and the CMRS Dual Brain Coil will be carried out according to the SOP's developed by the TBRRI and Xemed LLC.

MRI scanning will be performed with a MR Tech and Registered Respiratory Therapist present. Dispensing of 129Xe will be monitored using a gas dispensing form and a drug accountability log. This study will have a monitor assigned to it from the TBRRI that is not involved in this clinical trial. This is to ensure participant safety and adherence to the protocol.

ELIGIBILITY:
Inclusion Criteria:

A participant is eligible for inclusion in the study if the individual meets all of the following criteria:

1. Self-reported proficiency in English language.
2. Equal to or more than 8 years of education.
3. Normal or corrected to normal vision.
4. Able to provide informed consent.
5. Able to hold their breath for 20 seconds.

Normal cognition for healthy participant group inclusion criteria:

1. Preserved independence in functional abilities.
2. MoCA score no less than 26.
3. Males and non-lactating females of 18 to 85 years of age.

Alzheimer's disease group inclusion criteria:

1. Participants meet National Institute on Aging-Alzheimer's Association for probable or possible Alzheimer's Disease dementia.
2. MoCA score no less than 16.
3. Males and non-lactating females of 60 to 85 years of age.
4. Have a family member, close friend, or LAR that can be present for the informed consent process and study visits.

Exclusion Criteria:

A participant is ineligible for the study if the individual meets any of the following criteria:

1. Serious underlying medical condition, other, then the condition being investigated, which may affect cognitive function of the participant (in the opinion of the investigator): substance abuse, psychotic or depressive disorder, advanced or poorly controlled cardiac, pulmonary, hepatic, renal, neurological disorders in which the patient has significant speech, visual, motor or cognitive deficit, seizure disorders, endocrine or infectious disease or active malignancy.
2. MRI incompatibility as determined by MR Technologist during MRI screening.
3. Self-identifies as claustrophobic.
4. Female exclusion only: Are or may be pregnant; Planning on becoming pregnant.
5. Is a student currently enrolled in a course at Lakehead University where the Principal Investigator (PI) is the instructor.
6. Is a student currently enrolled in a degree program at Lakehead University where the PI is their direct thesis supervisor.
7. Is currently an employee of the PI at the Thunder Bay Regional Research Institute (TBRRI) and/or Lakehead University.

Normal cognition group exclusion criteria:

1. History of diagnosed neurological disease or injury.

Alzheimer's disease group exclusion criteria:

1. Existing diagnosis of dementia of etiology other than Alzheimer's disease.
2. Acute Delirium on the day of scanning (CAM tool assessment)

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2016-06-27 (Actual); Primary Completion 2022-04-19 (Actual); Study Completion 2022-04-19 (Actual)

PRIMARY OUTCOMES:
Signal-to-Noise Ratio (SNR) | Three years
  All scans will be optimized for the highest SNR possible; No aggregation of data

SECONDARY OUTCOMES:
P-Value | Three years
  To be calculated from a students paired t-test for signal change between healthy participant scans and participants with Alzheimer disease

CONTACTS AND LOCATIONS:
Overall Officials: Mitchell Albert, Ph.D., Principal Investigator — Thunder Bay Regional Health Research Institute
Locations (1):
- Thunder Bay Regional Health Sciences Centre, Thunder Bay, Ontario, Canada

REFERENCES:
- [Background] Agosta F, Pievani M, Geroldi C, Copetti M, Frisoni GB, Filippi M. Resting state fMRI in Alzheimer's disease: beyond the default mode network. Neurobiol Aging. 2012 Aug;33(8):1564-78. doi: 10.1016/j.neurobiolaging.2011.06.007. Epub 2011 Aug 3. PMID 21813210
- [Background] Albert MS, Cates GD, Driehuys B, Happer W, Saam B, Springer CS Jr, Wishnia A. Biological magnetic resonance imaging using laser-polarized 129Xe. Nature. 1994 Jul 21;370(6486):199-201. doi: 10.1038/370199a0. PMID 8028666
- [Result] Hane FT, Li T, Plata JA, Hassan A, Granberg K, Albert MS. Inhaled Xenon Washout as a Biomarker of Alzheimer's Disease. Diagnostics (Basel). 2018 Jun 6;8(2):41. doi: 10.3390/diagnostics8020041. PMID 29882765
- [Result] Grynko V, Shepelytskyi Y, Li T, Hassan A, Granberg K, Albert MS. Hyperpolarized 129 Xe multi-slice imaging of the human brain using a 3D gradient echo pulse sequence. Magn Reson Med. 2021 Dec;86(6):3175-3181. doi: 10.1002/mrm.28932. Epub 2021 Jul 17. PMID 34272774
- [Result] Shepelytskyi Y, Grynko V, Rao MR, Li T, Agostino M, Wild JM, Albert MS. Hyperpolarized 129 Xe imaging of the brain: Achievements and future challenges. Magn Reson Med. 2022 Jul;88(1):83-105. doi: 10.1002/mrm.29200. Epub 2022 Mar 7. PMID 35253919
- [Result] Shepelytskyi Y, Grynko V, Li T, Hassan A, Granberg K, Albert MS. The effects of an initial depolarization pulse on dissolved phase hyperpolarized 129 Xe brain MRI. Magn Reson Med. 2021 Dec;86(6):3147-3155. doi: 10.1002/mrm.28918. Epub 2021 Jul 13. PMID 34254356
- [Result] Shepelytskyi Y, Hane FT, Grynko V, Li T, Hassan A, Albert MS. Hyperpolarized 129Xe Time-of-Flight MR Imaging of Perfusion and Brain Function. Diagnostics (Basel). 2020 Aug 25;10(9):630. doi: 10.3390/diagnostics10090630. PMID 32854196